CLINICAL TRIAL: NCT05609500
Title: Warfarin Dosage Adjustment for Outside Therapeutic Range: a Linear Regression Model Analysis
Brief Title: Warfarin Dosage Adjustment Model Analysis Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Professor Bryan Ping Yen YAN (byan) (Unknown)
Responsible Party: Principal Investigator, Gormin Tan, Assistant professor, Chinese University of Hong Kong
Other Study IDs: 2022.370
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Warfarin
Keywords: Warfarin; dosage adjustment; therapeutic range; linear regression model

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Warfarin dosage adjustment model — Warfarin dosage adjustment model use to predict the initiation and the maintenance dose of warfarin. Variation of warfarin dose during stable maintenance phase for the same patient might be influenced more by temporal factors such as modification of drug regimens that utilize the CYP450 pathway, or dietary vitamin K intake

SUMMARY:
Despite the wide availability of Direct oral anticoagulation (DOAC), warfarin remains an important oral anticoagulant1 especially in patients with mechanical valve replacement or chronic renal failure where the evidence of DOAC is limited. However, the dosing of warfarin is challenging as it has a narrow therapeutic index and is highly influenced by dietary vitamin K intake and drugs that interacts with cytochrome (CYP) P4501. The time outside therapeutic range will carry the risk of adverse events such as thrombosis and bleeding. Numerous algorithms have been proposed that utilized either clinical or pharmacogenetics factors. The Clinical Pharmacogenetics Implementation Consortium (CPIC) has recommended the use of 4 dosing algorithms. However, these algorithms require the input of genetic information such as CYP2C9 and VKORC1 type which are not widely available locally and are less relevant in maintenance phase. Furthermore, these algorithms target mainly at predicting the initiation and the maintenance dose of warfarin. This has provided us with the opportunities to explore the Prediction model for on-treatment warfarin dose titration for outside therapeutic range.

DETAILED DESCRIPTION:
Despite the wide availability of Direct oral anticoagulation (DOAC), warfarin remains an important oral anticoagulant1 especially in patients with mechanical valve replacement or chronic renal failure where the evidence of DOAC is limited. However, the dosing of warfarin is challenging as it has a narrow therapeutic index and is highly influenced by dietary vitamin K intake and drugs that interacts with cytochrome (CYP) P4501. The time outside therapeutic range will carry the risk of adverse events such as thrombosis and bleeding. Numerous algorithms have been proposed that utilized either clinical or pharmacogenetics factors. The Clinical Pharmacogenetics Implementation Consortium (CPIC) has recommended the use of 4 dosing algorithms. However, these algorithms require the input of genetic information such as CYP2C9 and VKORC1 type which are not widely available locally and are less relevant in maintenance phase. Furthermore, these algorithms target mainly at predicting the initiation and the maintenance dose of warfarin. This has provided us with the opportunities to explore the Prediction model for on-treatment warfarin dose titration for outside therapeutic range.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been on maintenance warfarin treatment
2. Patients whose INR have fallen outside therapeutic range will be identified using CDARS enquiry

Exclusion Criteria:

1. No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is based on the primary objective, previous data in Hong Kong and calculation
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-09-06 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
extreme outside therapeutic range | 1 year
  INR<1.5 or INR>3.5 on two consecutive blood checking

SECONDARY OUTCOMES:
the time needed to achieve within therapeutic range | 1 year
  It is calculated by the time interval from the outside therapeutic range INR to final within therapeutic range INR, the number of INRs checking between the initial outside therapeutic range and the final within therapeutic range

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Yan, Study Chair — Chinese University of Hong Kong; Guangming Tan, Study Chair — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Johnson JA, Caudle KE, Gong L, Whirl-Carrillo M, Stein CM, Scott SA, Lee MT, Gage BF, Kimmel SE, Perera MA, Anderson JL, Pirmohamed M, Klein TE, Limdi NA, Cavallari LH, Wadelius M. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for Pharmacogenetics-Guided Warfarin Dosing: 2017 Update. Clin Pharmacol Ther. 2017 Sep;102(3):397-404. doi: 10.1002/cpt.668. Epub 2017 Apr 4. PMID 28198005
- [Background] Pokorney SD, Simon DN, Thomas L, Fonarow GC, Kowey PR, Chang P, Singer DE, Ansell J, Blanco RG, Gersh B, Mahaffey KW, Hylek EM, Go AS, Piccini JP, Peterson ED; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) Investigators. Patients' time in therapeutic range on warfarin among US patients with atrial fibrillation: Results from ORBIT-AF registry. Am Heart J. 2015 Jul;170(1):141-8, 148.e1. doi: 10.1016/j.ahj.2015.03.017. Epub 2015 Apr 1. PMID 26093875
- [Background] International Warfarin Pharmacogenetics Consortium; Klein TE, Altman RB, Eriksson N, Gage BF, Kimmel SE, Lee MT, Limdi NA, Page D, Roden DM, Wagner MJ, Caldwell MD, Johnson JA. Estimation of the warfarin dose with clinical and pharmacogenetic data. N Engl J Med. 2009 Feb 19;360(8):753-64. doi: 10.1056/NEJMoa0809329. PMID 19228618
- [Background] Sconce EA, Khan TI, Wynne HA, Avery P, Monkhouse L, King BP, Wood P, Kesteven P, Daly AK, Kamali F. The impact of CYP2C9 and VKORC1 genetic polymorphism and patient characteristics upon warfarin dose requirements: proposal for a new dosing regimen. Blood. 2005 Oct 1;106(7):2329-33. doi: 10.1182/blood-2005-03-1108. Epub 2005 Jun 9. PMID 15947090
- [Background] Gage BF, Eby C, Johnson JA, Deych E, Rieder MJ, Ridker PM, Milligan PE, Grice G, Lenzini P, Rettie AE, Aquilante CL, Grosso L, Marsh S, Langaee T, Farnett LE, Voora D, Veenstra DL, Glynn RJ, Barrett A, McLeod HL. Use of pharmacogenetic and clinical factors to predict the therapeutic dose of warfarin. Clin Pharmacol Ther. 2008 Sep;84(3):326-31. doi: 10.1038/clpt.2008.10. Epub 2008 Feb 27. PMID 18305455
- [Background] Anderson JL, Horne BD, Stevens SM, Grove AS, Barton S, Nicholas ZP, Kahn SF, May HT, Samuelson KM, Muhlestein JB, Carlquist JF; Couma-Gen Investigators. Randomized trial of genotype-guided versus standard warfarin dosing in patients initiating oral anticoagulation. Circulation. 2007 Nov 27;116(22):2563-70. doi: 10.1161/CIRCULATIONAHA.107.737312. Epub 2007 Nov 7. PMID 17989110
- [Background] Lenzini P, Wadelius M, Kimmel S, Anderson JL, Jorgensen AL, Pirmohamed M, Caldwell MD, Limdi N, Burmester JK, Dowd MB, Angchaisuksiri P, Bass AR, Chen J, Eriksson N, Rane A, Lindh JD, Carlquist JF, Horne BD, Grice G, Milligan PE, Eby C, Shin J, Kim H, Kurnik D, Stein CM, McMillin G, Pendleton RC, Berg RL, Deloukas P, Gage BF. Integration of genetic, clinical, and INR data to refine warfarin dosing. Clin Pharmacol Ther. 2010 May;87(5):572-8. doi: 10.1038/clpt.2010.13. Epub 2010 Apr 7. PMID 20375999